CLINICAL TRIAL: NCT06379451
Title: An Exploratory Clinical Study of the Safety and Efficacy of NKG2D Chimeric Antigen Receptor NK Cell Injections for the Treatment of Efractory Recurrent Multiple Myeloma
Brief Title: An Clinical Study of NKG2D-CAR-NK Cells for the Treatment of Refractory Recurrent Multiple Myeloma
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Changzhou No.2 People's Hospital (Other)
Responsible Party: Principal Investigator, Lu Xuzhang, Director of Hematology Department, Changzhou No.2 People's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2023]YLJSA088
Record Dates: First submitted 2024-04-17; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose group (Experimental): CAR-NK cell count 6x10^8
  Interventions: Drug: NKG2D Chimeric Antigen Receptor NK Cell Injection
- Medium dose group (Experimental): CAR-NK cell count 1x10^9
  Interventions: Drug: NKG2D Chimeric Antigen Receptor NK Cell Injection
- High dose group (Experimental): CAR-NK cell count 1.5x10^9
  Interventions: Drug: NKG2D Chimeric Antigen Receptor NK Cell Injection

INTERVENTIONS:
Drug: NKG2D Chimeric Antigen Receptor NK Cell Injection — Administer KN1102 cell injection three times on day 0, day 7, and day 14, respectively.
  Other Names: KN1102 cell injection

SUMMARY:
Multiple myeloma (MM) is a malignant disease characterized by the abnormal proliferation of clonal plasma cells. However, multiple myeloma remains an incurable disease and requires the exploration of more effective treatment methods to improve the efficacy of relapsed refractory multiple myeloma and prolong survival time.Currently, clinical application of CAR-T is mostly based on autologous T cell preparation, while relapsed/refractory AML patients have undergone multiple chemotherapy treatments, resulting in impaired self-T cell function, which affects the efficacy and prognosis of CAR-T therapy. Therefore, it is necessary to find new alternative treatments. NK cells are important immune cells in the body and are an important component of innate immunity. Compared with CAR-T cell therapy, CAR-NK cells have unique advantages in adoptive cell therapy. NKG2D receptor is an activating receptor expressed on NK cells, which can recognize NKG2D ligands (NKG2DL) expressed on tumor cells, activating NK cell killing activity through NKG2D-NKG2DL interaction. Therefore, the investigators plan to treat relapsed multiple myeloma by infusing NKG2D-CAR-NK cells to evaluate its efficacy and safety.

DETAILED DESCRIPTION:
Multiple Myeloma (MM) is a malignant disease with clonal abnormal plasma cell proliferation. It is the second most common malignant tumor in hematological system tumors. The incidence rate is 2-3/100000, and it is still incurable. In recent years, with the application of new drug based regimens such as proteasome inhibitors, immunomodulators, and anti CD38 monoclonal antibodies, the remission rate of MM patients has been significantly improved and chemotherapy related toxic side effects have been reduced, increasing the survival period of multiple myeloma from 2-3 years to more than 5 years. Sequential autologous hematopoietic stem cell transplantation after intensified induction therapy is currently the preferred treatment strategy for patients suitable for hematopoietic stem cell transplantation. For relapsed refractory MM, new generation oral proteasome inhibitors, monoclonal antibodies, and specific cellular immunotherapy have shown good therapeutic effects. However, multiple myeloma is still an incurable disease, and more effective treatment methods need to be explored to improve the efficacy and prolong survival time of relapsed and refractory multiple myeloma.

In recent years, CAR-T has achieved significant therapeutic effects in hematological malignancies. Chimeric antigen receptor T cell (CAR-T) immunotherapy is a rapidly developing new approach to tumor adoptive immunotherapy in recent years. Its main feature is to obtain T cells that recognize tumor antigen-specific receptors through genetic engineering modification, and endow them with targeting, killing, and persistence. CAR-T studies with MM antigen specificity have also been carried out and achieved good results. CAR-T cell therapy has become an effective new treatment for MM, with B-cell mature antigen (BCMA) becoming a clear target for CAR-T cell therapy. BCMA CAR-T cells can recognize and kill MM cells derived from MM patients, and exert anti-tumor effects in MM model mice through the perforin pathway. The overall effective rate of anti mouse derived BCMA CAR-T cell therapy for recurrent/refractory MM can reach 81%, with a CR rate of 55.5% for patients and a strict complete remission (sCR) of 13.3%. However, as the application time of CART cell therapy increases, recurrence remains an unavoidable issue, with approximately 40% of patients receiving CR still experiencing recurrence. Meanwhile, studies have shown that multi target CAR-T may prolong the remission period and reduce recurrence. Expanding the coverage of MM cell targets and clearing poorly differentiated MM cells may further improve the efficacy of CAR-T in treating relapsed refractory MM. Studies in mouse experimental models have confirmed that the combination of anti-CS1 CAR-T and anti-BCMA CAR-T has better therapeutic effects on myeloma cells than using anti-BCMA CAR-T alone. Clinical trials have confirmed the use of mouse derived anti BCMA CAR-T cells combined with humanized anti CD19 CAR-T cell infusion for the treatment of relapsed and refractory MM, with an ORR of 95.2% and a negative MRD conversion rate of 81.0%. However, with the extension of follow-up time, patients gradually experience recurrence. Therefore, although CAR-T therapy has shown positive clinical results in the treatment of multiple myeloma, recurrence remains a difficult problem to overcome, and more treatment methods are needed to address this issue.

Although CAR-T cells have strong tumor killing ability and specific targeted binding, the problems in CAR-T therapy cannot be ignored. Firstly, CAR-T therapy has related toxic side effects, mainly including: (1) Autoimmune toxicity mainly refers to the "on target/off tumor" toxic reaction. CAR cells attack tumor cells while also attacking normal tissues expressing the same antigen, causing damage to normal tissues. (2) Cells Factor release syndrome (CRS), which is a non antigen-specific toxicity caused by high levels of immune activation beyond the physiological state, is also the most prominent toxic response of CAR-T cell immunotherapy. CRS is often accompanied by an increase in various inflammatory cytokines, such as IL-2, IL-6, IL-10, TNF-a, and IFN- γ Wait. The clinical manifestations of CRS vary greatly, with fever being the most common, muscle pain, nausea, unstable hypotension, and hypoxia frequently occurring. The overall symptoms can range from mild flu like symptoms to severe life-threatening symptoms such as respiratory distress, multiple organ dysfunction, and even failure. (3) Neurotoxicity also appeared in some subjects, which is an unexpected toxic side effect that mainly includes symptoms such as blurred consciousness, coma, aphasia, motor disorders, and seizures. Secondly, the preparation cycle of CAR-T cells is long and not suitable for patients with rapid disease progression. At present, the preparation of CAR-T cells in the study population is mostly based on autologous peripheral blood collection and lentivirus transfection. T cells need to undergo a series of operations such as sorting, activation, transfection, and amplification before being reintroduced to patients, which generally takes 2-3 weeks. On the one hand, it cannot meet the urgent treatment needs of patients with rapid disease progression, and on the other hand, long-term in vitro cultivation leads to excessive differentiation of CAR-T cells in vivo, resulting in reduced survival, proliferation, and killing ability in vivo, reducing therapeutic efficacy. Finally, the efficacy of CAR-T may be affected by early chemotherapy. At present, the clinical application of CAR-T is mostly prepared by autologous T cells, and patients with relapsed/refractory AML have received multiple chemotherapy treatments, resulting in impaired T cell function, which affects the efficacy of CAR-T and patient prognosis. Therefore, it is necessary to seek new alternative treatments.

NK cells are important immune cells in the body and an important component of innate immunity. Under physiological conditions, NK cell inhibitory receptors recognize MHC class I molecules widely expressed on the surface of normal tissue cells, which inhibits NK cell function and prevents them from killing their own normal tissue cells. In tumor tissue, due to the downregulation of MHC class I molecule expression on the surface of tumor cells, ligands that activate receptors such as NKp30, NKp44, NKp46 are upregulated, leading to NK cell activation and ultimately killing tumor cells. CAR-NK cells express CAR molecules on the surface of NK cells, recognize target antigens through CAR, and further activate NK cells to kill tumor cells. The CAR structure of CAR-NK cells usually consists of three parts, namely the extracellular antigen binding domain, transmembrane domain, and intracellular activation domain, which is very similar to the CAR structure used in CAR-T cell therapy. According to the different intracellular domains, CAR structures will also be compared and validated accordingly.

Compared to CAR-T cell therapy, CAR-NK cells have their unique advantages in adoptive cell therapy: 1) The probability of CAR-NK cells experiencing cytokine storms is low. The pro-inflammatory cytokines secreted by CAR-T cells, such as IL-1 and IL-6, are the main cytokines causing CRS. Active CAR-NK cells typically produce TNF- α There is a significant difference between the types of cytokines produced by granulocyte macrophage colony-stimulating factor (GM-CSF) and T lymphocytes. Clinical studies have shown that CAR-NK treatment significantly reduces the probability of cytokine storms. 2) CAR-NK cells have multiple killing mechanisms that can kill tumor cells with low or no expression of target antigens, reducing the recurrence of target antigen negative tumors. CAR-T cells are difficult to recognize target cells with low or no expression of target antigens, and these cells cannot be cleared, leading to tumor recurrence. CAR-NK cells not only recognize tumor surface antigens through single chain antibodies to kill tumor cells, but also activate various receptor recognition ligands to kill tumor cells. Such as natural cytotoxic receptors (NKp46, NKp44, and NKp30), NKG2D, and DNAM-1. In addition, NK cells pass through Fc γ RIII (CD16) induces antibody dependent cytotoxicity, and multiple mechanisms combine to kill heterogeneous tumor cells, thereby reducing the risk of tumor recurrence. 3) Allogeneic transplantation of CAR-NK cells does not cause graft-versus-host disease (GvHD). When CAR-T cells in the test population are generated by healthy donors who do not match human leukocyte antigen (HLA), Non autogenous MHCs expressed on allogeneic CAR-T cells can induce immune rejection and cause severe hematological toxicity. NK cells are innate immune cells that do not rely on MHCs molecular recognition. Allogeneic CAR-NK cells do not induce GvHD production. 4) NK cells come from multiple sources to meet the needs of patients whose cell quality and quantity are affected by multiple chemotherapy treatments. NK cells can be obtained from human umbilical cord blood, peripheral blood, induced pluripotent stem cells, and NK-92 cell lines. For patients who have difficulty collecting sufficient cells due to multiple chemotherapy treatments, multiple sources of NK cells can meet the needs of CAR-NK treatment. 5) CAR-NK cells can provide timely "spot type" treatment. NK cells are not limited by major histocompatibility complexes, therefore, allogeneic NK cells can be used for modification and development into off the shelf CAR-NK cell therapy. For patients with rapid tumor progression, timely treatment can be provided to avoid disease progression due to waiting for cell preparation.

The NKG2D receptor is an activating receptor that expresses NK cell expression. It can recognize the NKG2D ligand (NKG2DL) expressed in tumor cells and activate NK cell killing activity through NKG2D-NKG2DL interactions. NKG2DL is located at different positions on chromosome 6 and belongs to two gene families, including MICA/MICB and ULBPs. The NKG2D ligand is expressed at different levels on the surface of tumor cells or virus infected cells, while it is not expressed on the surface of normal cells, with over 70% of human tumor cells showing upregulation of the NKG2D ligand. Our previous research has shown that the U266 myeloma cell line and over 62% of MM patients express different levels of NKG2D ligands, and immune cells can mediate the killing of MM cells through the interaction between NKG2D receptors and ligands. Targeted NKG2DL CAR-NK cell therapy for MM achieved good therapeutic effects in preclinical experiments. At the same time, 5 recurrent MM received NKG2D-CAR-NK cells without treatment-related adverse reactions, dose limiting toxicity, and no CRS response observed. A preclinical study has shown that NKG2D-CAR-NK has a more cytotoxic effect on MM cells than simply expanded and activated NK cells, providing a basis for the treatment of MM with NKG2D-CRA-NK.

Therefore, choosing NKG2DL as the target for treating AML has three main advantages: on the one hand, its specific expression on tumor cells can ensure the safety of CAR-NK drugs and avoid serious off target toxicity; In addition, the diversity of NKG2D ligands can to some extent avoid tumor recurrence caused by MM cell heterogeneity or single target deficiency, and better maintain drug efficacy; Finally, NKG2DL as a therapeutic target for MM has obtained positive clinical data. Therefore, the investigators plan to evaluate the efficacy and safety of combined infusion of NKG2D-CAR-NK cells in the treatment of recurrent multiple myeloma. The clinical data of this study can provide data support for new treatment plans for relapsed refractory MM.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 18 to 70 years old;
2. Expected survival time>12 weeks;
3. Diagnosed as multiple myeloma through physical examination, pathological examination, laboratory examination, and imaging;
4. Difficult to treat multiple myeloma patients;
5. Patients with recurrent multiple myeloma;
6. ALT, AST<3 times normal; Bilirubin<2.0mg/dl;
7. Quality of Life Score (KPS)>50%;
8. The patient has no serious diseases such as heart, liver, or kidney;
9. Recurrence or no remission of the disease after hematopoietic stem cell transplantation or cellular immunotherapy;
10. Inappropriate conditions for stem cell transplantation or abandonment of transplantation due to limitations in conditions;
11. Blood can be taken intravenously without any other contraindications for leukocyte removal surgery;
12. Can understand and voluntarily sign a written informed consent form.

Exclusion Criteria:

1. Pregnant or lactating women, or women with pregnancy plans within six months;
2. Infectious diseases (such as HIV, active tuberculosis, etc.);
3. Active hepatitis B or hepatitis C infection;
4. Feasibility assessment screening proves that the transfection of targeted lymphocytes is less than 10% or the amplification is insufficient (<5-fold) under the co stimulation of CD3/CD28;
5. Abnormal vital signs and inability to cooperate with the examination;
6. Individuals with mental or psychological disorders who cannot cooperate with treatment and efficacy evaluation;
7. Highly allergic constitution or a history of severe allergies, especially those who are allergic to IL-2;
8. Subjects with systemic or severe local infections requiring anti infection treatment;
9. Subjects with severe autoimmune diseases;
10. The doctor believes that there are other reasons why patients cannot be included in treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-04-18 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicity (DLTs) | within 4 weeks after infusion; 12, 24, 36 and 52 weeks after infusion
  To characterize the Dose Limiting Toxicities (DLTs) of NKG2D-CAR-NK Cells for refractory recurrent multiple myeloma
Treatment Emergent Adverse Events (TEAEs) | within 4 weeks after infusion; 12, 24, 36 and 52 weeks after infusion
  To characterize the Treatment Emergent Adverse Events (TEAEs) of NKG2D-CAR-NK Cells for refractory recurrent multiple myeloma

SECONDARY OUTCOMES:
Objective Response Rate of subjects | Time Frame: 2, 4, 8, 12, 16, 24, 28, 40 and 52 weeks after first infusion
  The target response is evaluated according to the definition of the International MM Working Group. Objective response rate is defined as having bone marrow morphology and immune classification

CONTACTS AND LOCATIONS:
Overall Officials: Xuzhang Lu, doctor, Study Director — The Second People's Hospital of Changzhou; Liming Tang, doctor, Study Chair — The Second People's Hospital of Changzhou
Locations (1):
- Changzhou Second People's Hospital, Changzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
publish one's thesis